CLINICAL TRIAL: NCT03879434
Title: Routine Application of Ostenil® Mini in Patients with Rhizarthrosis
Status: Completed | Type: Observational
Sponsor: TRB Chemedica AG (Industry)
Responsible Party: Sponsor
Other Study IDs: OSTCMC-PMCF-DE-2018-01
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Rhizarthrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ostenil® Mini: 1-3 injections of sodium hyaluronate 1.0 % (10 milligrams (mg) / 1,0 millilitres (ml)) in weekly interval.
  Interventions: Device: Ostenil® Mini

INTERVENTIONS:
Device: Ostenil® Mini — Ostenil® Mini is a CE-certified viscoelastic solution for injection into the Joint cavity, containing 1.0 % sodium hyaluronate from fermentation

SUMMARY:
PMCF study to observe the routine application of Ostenil® Mini in the treatment of pain and restricted mobility in degenerative and traumatic changes of the CMC joint.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years of age and in good general health condition
* Signed informed consent
* Existing Ostenil® Mini recommendation for the treatment of rhizarthrosis

Exclusion Criteria:

* Known hypersensitivity to one of the Ostenil® Mini components
* Known pregnancy or lactating females
* Presence of coagulation disorder
* Subjects not capable of contracting and of understanding the nature, risks, significance and implications of the clinical investigation and unable to form a rational intention in the light of these facts
* Subjects unable to understand informed consent or having a high probability of non compliance to the study procedures and / or non completion of the study according to investigator's judgement (e.g. illiteracy, insufficient knowledge of local language)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with Rhizarthrosis and a Recommendation for Treatment with Ostenil® Mini.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Change of Pain Intensity compared to Baseline (VAS-slider) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Evaluation of Pain Intensity by the Patient on a 10 cm VAS-slider. (10 cm equal the worst pain)
Change of Subjective Therapy Evaluation (FIHOA Questionnaire, 4 grade scale) compared to Baseline | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Functional Index for Hand OsteoArthritis (FIHOA) to assess hand-OA related functional impairment on a 4-grade scale
Change of Subjective Quality of Life Evaluation (Questionnaire with 5 Point Likert scale) compared to Baseline | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Questionnaire to assess hand-OA related Quality of Life on a 5-grade scale
Change of Subjective Symptom Evaluation (Overall Impression on a scale from 1 to 5) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  The Change of Overall Subjective Symptom Evaluation on a scale from 1 (much improved) to 5 (much worse)
Incidence of Treatment-Emergent Adverse Events | Up to Day 252 after the last injection
Change of Key Pinch Strength compared to Baseline (Pinch Gauge) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Measurement of Key Pinch in kilograms with a Pinch Gauge
Change of Tip Pinch Strength compared to Baseline (Pinch Gauge) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Measurement of Tip Pinch in kilograms with a Pinch Gauge
Change of Palmar Pinch Strength compared to Baseline (Pinch Gauge) | Day 7, Day 14, Day 84 after last injection, Day 168 after last injection
  Measurement of Palmar Pinch in kilograms with a Pinch Gauge

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Orthopädie am Tauentzien, Berlin, State of Berlin
  - Praxis für Orthopädie und Unfallchirurgie, Berlin
  - MVZ Berlin Freiheit 1, Berlin
  - Orthopädie am Kiesteich, Berlin
  - Wirbelsäulen Gelenk Zentrum Westend, Berlin
  - Orthopädie Wannsee, Berlin